CLINICAL TRIAL: NCT05518318
Title: Evaluate the Efficacy and Safety of GLS-010 Versus Chemotherapy Assessed by Investigator in Patients With Relapsed or Refractory Classical Hodgkin's Lymphoma (R/R cHL) in a Randomized, Open, Multicenter Phase III Trial
Brief Title: GLS-010 Monotherapy Versus Chemotherapy in Patients With Relapsed or Refractory Classical Hodgkin's Lymphoma (R/R cHL)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Gloria Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLS-010-31
Record Dates: First submitted 2022-08-19; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Classic Hodgkin's Lymphoma; Recurrent Classic Hodgkin Lymphoma; Refractory Classic Hodgkin Lymphoma
Keywords: GLS-010; relapsed or refractory classic Hodgkin's lymphoma
MeSH Terms: conditions — Recurrence | interventions — zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLS-010 (Experimental): GLS-010 therapy
  Interventions: Drug: GLS-010
- chemotherapy (Active Comparator): chemotherapy
  Interventions: Drug: Chemotherapy of Investigator's choice

INTERVENTIONS:
Drug: GLS-010 — Participants receive GLS-010 240mg intravenously (IV) on Day 1, Q2W
  Other Names: GLS-010 therapy
  Arms: GLS-010
Drug: Chemotherapy of Investigator's choice — Chemotherapy administered as assessed as appropriate by the investigator in accordance with the local guideline, including but not limited to DHAP,GEMOX, ESHAP , ICE , IGEV and GVD
  Arms: chemotherapy

SUMMARY:
The primary objective of this study is to evaluate the efficacy of GLS-010 in participants with relapsed or refractory classical Hodgkin lymphoma (R/R cHL), as measured by Progression-free Survival (PFS) as assessed by IRRC

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed written informed consent form (ICF).
2. Age of ≥ 18 years at the time of enrollment.
3. Histologically confirmed classic Hodgkin's lymphoma (cHL).
4. Subjects required Relapsed or refractory ,failure to at least 2 lines of prior systemic chemotherapy.
5. Patients who have failed prior vibutuximab treatment or are unwilling or not eligible for vibutuximab treatment
6. Have at least one measurable lesion according to Lugano classification 2014 and FDG-PET was positive.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Life expectancy of ≥ 12 weeks.
9. Have adequate hematologic and organ function .

Key Exclusion Criteria:

1. Nodular lymphocytes are non-Hodgkin's lymphoma or gray area lymphoma.
2. Central nervous system lymphoma invasion.
3. Subjects requiring systemic corticosteroids or other immunosuppressive agents within 14 days prior to screening or during the study period.
4. Prior exposure to any anti-PD-1, anti-PD-L1,anti-PD-L2, anti-CD137,anti-CTLA-4 antibody, or any other antibody or drug target for T cell co-stimulatory or checkpoint pathways.
5. Known human immunodeficiency virus (HIV), or serologic status reflecting active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
6. Subjects with other malignancy within 5 years prior to the first dose of study treatment, except for Cervical carcinoma in situ and Cured basal cell carcinoma of the skin.
7. Have received chemotherapy, radiotherapy, molecular-targeted therapy or major surgery within 4 weeks prior to the first dose of study treatmen; Clinically significant AE associated with previous treatment has not returned to baseline or ≤1 (except hair loss).
8. Pregnant or breast-feeding women.
9. Patients are unsuitable for the study evaluated by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by Independent Radiologic Review Committee (IRRC) per Lugano Classification 2014 | Up to 2 years
  Time from the date of randomization to the date of progressive disease (PD) or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 2 years
  Defined as the time from the date of randomization to the date of death due to any Defined as the time from the date of randomization to the date of death due to any reason
Objective Response Rate (ORR) | Up to 2 years
  ORR defined as the proportion of subjects who achieves a best overall response of CR or PR based on Lugano 2014 classification.
Disease Control Rate (DCR) | Up to 2 years
  DCR defined as the proportion of subjects' response of CR, PR, or SD based on Lugano Classification 2014.
Duration of Response (DoR) | DoR defined as the time from the date that CR or PR are first occurred to the date of objective disease progression or death, whichever occurs first
  Up to 2 years
Time to Response (TTR) | TTR defined as the time from the date of randomization to the date when the response criteria are first met, based on Lugano Classification 2014
  Up to 2 years

OTHER OUTCOMES:
Number of subjects with adverse events (AEs) | From the time of signed informed consent through 90 days after the last dose of GLS-010
  Up to 2 years